CLINICAL TRIAL: NCT05228561
Title: The Effect of Mobile Application Supported Diabetes Education On Type 2 Diabetes Self-Management And Blood Sugar In Newly Diagnosed Type 2 Diabetes Patients
Brief Title: The Effect of Mobile Application Supported Diabetes Education On Type 2 Diabetes Self-Management And Blood Sugar Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, EMRE TURHAN, Graduate Student, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EgeUniversity-ETURHAN-001
Record Dates: First submitted 2021-12-30; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 2; Education; Mobile Applications; Self-Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): After the physician involved in the study asks the participants for their biochemical tests (FBC, HbA1C, LDL-C, HDL-C, Total K, Triglyceride), the outpatient dietitian will give routine nutrition education to the participants. In addition, a data collection form including socio-demographic information, health history, nutrition history and height, weight, waist circumference measurements will be made and filled by the thesis student.
- Study Group (Experimental): The software developed for this research will be downloaded to the phones of the participants in the intervention group. With this software prepared, written and visual information (pictures, mini-videos) will be given to participants every day for 3 months on diabetes, self-management of diabetes and nutrition. Whether the participants read the messages or not will also be monitored through this software. At the end of 3 months, the participants in the intervention and control groups will be invited again, and their biochemical parameters and self-management status will be measured according to the diabetes self-management scale. Data will be collected through face-to-face interviews in the outpatient clinic, and weight will be measured with the bioelectrical impedance analyzer in the outpatient clinic, height will be measured with a height meter fixed to the wall, and waist circumference will be measured with a non-stretchable measuring tape.
  Interventions: Other: Mobile Application Supported Nutrition and Diabetes Education

INTERVENTIONS:
Other: Mobile Application Supported Nutrition and Diabetes Education — With this intervention, the difference between the mobile application supported nutrition diabetes education created with written and visual (video) and face-to-face nutrition and diabetes education will be found.
  Arms: Study Group

SUMMARY:
Diabetes is one of the biggest public health problems of the 21st century. Type 2 diabetes mellitus accounts for more than 90% of all diabetes cases and is the most common type of diabetes. Type 2 diabetes, in which genetic and environmental factors play a role,It is a metabolic disorder in which insulin resistance, decrease in insulin secretion and incretin hormone deficiency are effective in its physiopathology, characterized by polydipsia, polyphagia and polyuria, where the organism cannot adequately benefit from carbohydrates, fats and proteins due to insulin deficiency or defects in the effect of insulin, which requires continuous medical care.

Diabetes is a major cause of blindness, end-stage renal disease, coronary artery disease, stroke and inferior extremity amputations. These complications due to diabetes impair the patient's quality of life and impose social, financial and emotional burdens on both the patient and their family.

Diabetes education should be provided by healthcare professionals in order to ensure that diabetes patients knowledge and skills to prevent complications and provide better self management and self-care.

However, The fact that individuals do not have time to spare for face-to-face health education, the possibility of accessing information in the web environment repeatedly and the lower cost of education in the web environment compared to classical education increases the importance of web-based health education. The widespread use of mobile technologies in recent years has led to the development of new mobile applications related to diabetes.

The disquisition proposal the investigators prepared was created to investigate the effect of mobile application supported diabetes and nutrition education on type 2 diabetes self-management and blood sugar in newly diagnosed type 2 diabetes patients.

In this context, with the development of a mobile application prepared in visual, text and video format to provide diabetes education, the monitoring of blood parameters before and after diabetes education, and the implementation of the Type 2 Diabetes Self-Management Scale, (which consists of 19 items developed in 2020), and type 2 diabetes self-management and the effect on blood sugar will be examined. This study will provide answers to questions about the effectiveness of diabetes education given to Type 2 Diabetes patients via mobile applications on diabetes self-management and blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes patients in the endocrinology and metabolism outpatient clinic of Ege University Medical Faculty Hospital.
* Patients with Type 2 DM, between the ages of 18-64, using smart phones and having regular internet will be included in the study.

Exclusion Criteria:

* Those who receive regular messages every day will be checked, and those who do not open/read more than 25% of the messages in total will be excluded.
* type 1 diabetes or gestational diabetes

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
The effect of mobile application supported diabetes education on type 2 diabetes self-management. | 6 Month
  Type 2 diabetes self-management scores of the participants in the study group and control group will be compared.
  For this comparison, the "Type 2 Diabetes Self-Management Scale" consisting of 3 sub-titles (Healthy Lifestyle Behaviors, Blood Sugar Management, Health Services Use) and 19 items developed in 2020 will be applied.
  (Scoring: Always 5, Often 4, Sometimes 3, Rarely 2, Never 1 point). Those with higher scores will be considered to show better self-management. This scale will first be administered to the participants when they are diagnosed with type 2 diabetes in the hospital.
  Participants will be given diabetes and nutrition education for 3 months, and the Type 2 Diabetes Self-Management Scale will be repeated by inviting them to the hospital for control.
  Then, the participants will be taken into a 3-month follow-up process and at the end of the process, they will be invited to the hospital for control and the Type 2 Diabetes Self-Management Scale will be repeated.
The effect of mobile application supported diabetes education on blood sugar | 6 Months
  The physician participating in the study will measure the Fasting Blood Sugar (mg/dl) values of the participants.
  When the participants are diagnosed with type 2 diabetes, their Fasting Blood Sugar (mg/dl) values will be measured and a 3-month diabetes education will be given. At the end of this diabetes training, the participants will be invited to the hospital for control and their Fasting Blood Sugar (mg/dl) values will be measured again.
  Then, the participants will be taken to the 3-month follow-up process and at the end of the process, the participants will be invited to the hospital for control and their Fasting Blood Sugar (mg/dl) values will be measured again.
  At the end of the research, the effects of mobile application supported diabetes education on fasting blood sugar (mg/dl) will be compared with the routine diabetes education given in the hospital.

REFERENCES:
- [Background] Zimmet P, Alberti KG, Magliano DJ, Bennett PH. Diabetes mellitus statistics on prevalence and mortality: facts and fallacies. Nat Rev Endocrinol. 2016 Oct;12(10):616-22. doi: 10.1038/nrendo.2016.105. Epub 2016 Jul 8. PMID 27388988
- [Background] Satman I, Yilmaz T, Sengul A, Salman S, Salman F, Uygur S, Bastar I, Tutuncu Y, Sargin M, Dinccag N, Karsidag K, Kalaca S, Ozcan C, King H. Population-based study of diabetes and risk characteristics in Turkey: results of the turkish diabetes epidemiology study (TURDEP). Diabetes Care. 2002 Sep;25(9):1551-6. doi: 10.2337/diacare.25.9.1551. PMID 12196426
- [Background] Satman I, Omer B, Tutuncu Y, Kalaca S, Gedik S, Dinccag N, Karsidag K, Genc S, Telci A, Canbaz B, Turker F, Yilmaz T, Cakir B, Tuomilehto J; TURDEP-II Study Group. Twelve-year trends in the prevalence and risk factors of diabetes and prediabetes in Turkish adults. Eur J Epidemiol. 2013 Feb;28(2):169-80. doi: 10.1007/s10654-013-9771-5. Epub 2013 Feb 14. PMID 23407904
- [Background] Sami W, Ansari T, Butt NS, Hamid MRA. Effect of diet on type 2 diabetes mellitus: A review. Int J Health Sci (Qassim). 2017 Apr-Jun;11(2):65-71. PMID 28539866
- [Background] Millar A, Cauch-Dudek K, Shah BR. The impact of diabetes education on blood glucose self-monitoring among older adults. J Eval Clin Pract. 2010 Aug;16(4):790-3. doi: 10.1111/j.1365-2753.2009.01195.x. Epub 2010 Jun 14. PMID 20557415
- [Background] Powers MA, Bardsley JK, Cypress M, Funnell MM, Harms D, Hess-Fischl A, Hooks B, Isaacs D, Mandel ED, Maryniuk MD, Norton A, Rinker J, Siminerio LM, Uelmen S. Diabetes Self-management Education and Support in Adults With Type 2 Diabetes: A Consensus Report of the American Diabetes Association, the Association of Diabetes Care & Education Specialists, the Academy of Nutrition and Dietetics, the American Academy of Family Physicians, the American Academy of PAs, the American Association of Nurse Practitioners, and the American Pharmacists Association. Diabetes Care. 2020 Jul;43(7):1636-1649. doi: 10.2337/dci20-0023. Epub 2020 Jun 8. No abstract available. PMID 32513817
- [Background] Chomutare T, Fernandez-Luque L, Arsand E, Hartvigsen G. Features of mobile diabetes applications: review of the literature and analysis of current applications compared against evidence-based guidelines. J Med Internet Res. 2011 Sep 22;13(3):e65. doi: 10.2196/jmir.1874. PMID 21979293
- [Background] El-Gayar O, Timsina P, Nawar N, Eid W. Mobile applications for diabetes self-management: status and potential. J Diabetes Sci Technol. 2013 Jan 1;7(1):247-62. doi: 10.1177/193229681300700130. PMID 23439183
- [Background] Kelly L, Jenkinson C, Morley D. Experiences of Using Web-Based and Mobile Technologies to Support Self-Management of Type 2 Diabetes: Qualitative Study. JMIR Diabetes. 2018 May 11;3(2):e9. doi: 10.2196/diabetes.9743. PMID 30291098
- [Background] Norris SL, Lau J, Smith SJ, Schmid CH, Engelgau MM. Self-management education for adults with type 2 diabetes: a meta-analysis of the effect on glycemic control. Diabetes Care. 2002 Jul;25(7):1159-71. doi: 10.2337/diacare.25.7.1159. PMID 12087014
- [Background] Calderon JL, Shaheen M, Hays RD, Fleming ES, Norris KC, Baker RS. Improving Diabetes Health Literacy by Animation. Diabetes Educ. 2014 May;40(3):361-372. doi: 10.1177/0145721714527518. Epub 2014 Mar 27. PMID 24676274
- [Background] Abrar EA, Yusuf S, Sjattar EL, Rachmawaty R. Development and evaluation educational videos of diabetic foot care in traditional languages to enhance knowledge of patients diagnosed with diabetes and risk for diabetic foot ulcers. Prim Care Diabetes. 2020 Apr;14(2):104-110. doi: 10.1016/j.pcd.2019.06.005. Epub 2019 Jul 13. PMID 31311727
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- See also: Diabetes Atlas-Tenth Edition — https://diabetesatlas.org/atlas/tenth-edition/